CLINICAL TRIAL: NCT06722703
Title: ESWL Vs Flexible Uretroscopy in Management of Upper Ureteric Stones a Prospective Randomized Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Taha Abdulrahim Bassery Bakhit, resident doctor at urology department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESWL vs FURS UUS
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stone Ureter
Keywords: upper ureteric stones; ESWL; flexible uretroscopy
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESWL group (Experimental): The surgical technique of shock wave lithotripsy
  Interventions: Procedure: shock wave lithotripsy
- FURS group (Experimental): Flexible ureteroscope lithotripsy
  Interventions: Procedure: Flexible ureteroscope lithotripsy

INTERVENTIONS:
Procedure: shock wave lithotripsy — Extracorporeal shock wave lithotripsy will be performed using a third-generation electromagnetic lithotripter The focal depth is 110 mm; the focal area is 7 mm (radial) and 45-50 mm (axial), and the focal pressure is 6-30 MPa). The procedure is performed in a supine or prone position without anesthesia. Stone localization and simultaneous real-time monitoring during the process will be performed by ultrasound). The shock frequency is 60-90 (shock waves/min). The total number of shock waves applied for one session is between 1500 and 2500 waves, or the session is stopped at a significant stone fragmentation is detected. The voltage applied per session ranged from 10 to 16 kV with stepwise power ramping strategy. All procedures in the SWL group are outpatient procedures.
  Arms: ESWL group
Procedure: Flexible ureteroscope lithotripsy — All F-URS cases will be performed by a single surgeon (HMI). A guidewire is placed in the upper urinary tract through a rigid cystoscope under fluoroscopic guidance. An 8-10 F dual lumen catheter is used to dilate the intramural ureter and to fix a second guidewire with hydrophilic coat. The 7.5 F flexible ureteroscope is passed into the upper urinary tract in a monorail fashion over the second wire. A holmium-YAG laser is used at an energy setting of 0.8-1 J and a rate of 10-15 Hz. A 200 µm laser fibre is used for delivering laser energy to the stones. A 2.2 F tipless nitinol basket is used to displace the stones from the lower pole to an upper pole calyx before disintegration. Adequate fragmentation is considered when fragments are smaller than the diameter of the guide wire. Stone fragments will be left for spontaneous passage. At the end of the procedure, the whole collecting system will be inspected for residual stones and a double pigtail ureteric stent will be left for 2 weeks t
  Arms: FURS group

SUMMARY:
This comparison between ESWL and flexible ureteroscopy aims to explore the efficacy, safety, and outcomes of these treatments for upper ureteric stones under 15 mm, focusing on stone-free rates, procedural risks, recovery times, and recurrence rates. A thorough understanding of these techniques is essential for optimizing patient outcomes and personalizing treatment strategies.

study aim to evaluate the effectiveness, safety, and cost of SWL compared to flexible uretroscopy in management patients with upper ureteric stone less than 15 mm in size

DETAILED DESCRIPTION:
The management of upper ureteric stones, particularly those less than 15 mm in size, has seen significant advancements with the development of minimally invasive techniques. Urolithiasis is a common condition, and selecting the most appropriate treatment is crucial for effective stone clearance and minimizing complications. Two widely used approaches in treating upper ureteric stones are Extracorporeal Shock Wave Lithotripsy (ESWL) and Flexible Ureteroscopy (FURS).

ESWL, a non-invasive procedure, uses focused shock waves to fragment the stone into smaller pieces that can be passed naturally through the urinary tract. Its non-invasiveness makes it an attractive option for many patients; however, its success is influenced by factors such as stone composition, location, and patient anatomy. In contrast, Flexible Ureteroscopy (FURS) is a minimally invasive endoscopic technique where a flexible ureteroscope is passed through the urinary tract to directly visualize and fragment the stone using a laser (usually a Holmium: YAG laser). This method allows for a more targeted approach and is often used when ESWL is less effective or contraindicated.

ESWL and FURS have distinct advantages and limitations, and the choice between them depends on factors including stone size, density, location, and patient-specific considerations such as body habitus and anatomical variations.

ELIGIBILITY:
Inclusion Criteria:

* patients age>18 years old. Stone site: upper ureteric stone. Stone side: unilateral stones Stone size: stones diameter up to 1cm Stone number: single or multiple Radio-opaque stone

Exclusion Criteria:

* patients with solitary kidney or only function kidney renal impairment present of distal obstruction pregnancy, current breast feeding. Bleeding tendency or anticoagulation. ipsilateral ureterolithiasis, Acute or chronic nephritis, or Renal tuberculosis aneurysm of the aorta or renal artery. inability to position the patient on the SWL table (eg, due to severe skeletal deformity or morbid obesity).

radiolucent stones that are not visible on ultrasound. severe metabolic disturbances (eg, cystinuria, primary hyperparathyroidism, or renal tubular acidosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The stone-free rate (SFR) | 1 month
  The stone-free rate (SFR) is defined as no evidence of clinically significant stone fragments (≥ 4 mm in size) in combination with a plain X-ray of the urinary tract (KUB) and urinary ultrasound one month after SWL or F-URS

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yuri P, Hariwibowo R, Soeroharjo I, Danarto R, Hendri AZ, Brodjonegoro SR, Rasyid N, Birowo P, Widyahening IS. Meta-analysis of Optimal Management of Lower Pole Stone of 10 - 20 mm: Flexible Ureteroscopy (FURS) versus Extracorporeal Shock Wave Lithotripsy (ESWL) versus Percutaneus Nephrolithotomy (PCNL). Acta Med Indones. 2018 Jan;50(1):18-25. PMID 29686172
- [Background] Jahrreiss V, Seitz C, Quhal F. Medical management of urolithiasis: Great efforts and limited progress. Asian J Urol. 2024 Apr;11(2):149-155. doi: 10.1016/j.ajur.2023.05.001. Epub 2023 Jun 29. PMID 38680579